CLINICAL TRIAL: NCT06389877
Title: A Phase 1/2 Dose-exploration and Dose-expansion Study to Evaluate the Safety and Efficacy of BEAM-302 in Adult Patients With Alpha-1 Antitrypsin Deficiency (AATD)-Associated Lung Disease and/or Liver Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of BEAM-302 in Adult Patients With Alpha-1 Antitrypsin Deficiency (AATD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTX-302-001
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-01

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BEAM-302 Drug Product (Experimental)
  Interventions: Drug: BEAM-302

INTERVENTIONS:
Drug: BEAM-302 — BEAM-302 is a lipid nanoparticle (LNP)-based therapy for the treatment of patients with AATD

SUMMARY:
This is a Phase 1/2, multicenter, open-label, dose-exploration (Phase 1) and dose-expansion (Phase 2) study to evaluate the safety, tolerability, PK/PD, and efficacy of BEAM-302 in adult patients with AATD-associated lung disease and/or liver disease and to determine the optimal biological dose (OBD).

ELIGIBILITY:
Part A:

Inclusion Criteria:

* Males or females 18 - 70 years of age inclusive at the time of consent.
* Diagnosis of AATD and homozygous for the PiZZ mutation (confirmed by genetic testing).
* Blood total AAT level <11 μM or equivalent protein in mg/dL.
* Patients receiving augmentation therapy in regions where augmentation is not SoC must be willing to washout augmentation therapy for at least 6 weeks prior to signing the ICF and for the length of the study (unless clinically indicated)
* A postbronchodilator FEV1 ≥40% of predicted and an FEV1/FVC <70% at screening. (PFTs obtained within 1 year of signing the ICF may be used for eligibility.)
* Evidence of emphysema on a historic CT scan or a DLCO ≤70% of the predicted value (corrected for hemoglobin) at screening. (PFTs obtained within 1 year of signing the ICF may be used for eligibility.)

Exclusion Criteria:

* Body mass index >30
* Lung or liver transplant or on waiting list for lung or liver transplant or status post lung volume reduction surgery.
* Clinical evidence of severe bronchiectasis as per the discretion of the investigator (eg, excessive sputum production or recurrent infections requiring antibiotic use [>4x/year]).
* Liver disease with any of the following:

  * FibroScan liver stiffness measurement ≥7.5 kilopascals (kPa). (For sites without access to FibroScan, APRI >0.5 can be used as a surrogate exclusion criterion [Yilmaz, 2011].
  * Known history of liver cirrhosis or complications of cirrhosis (eg, varices, ascites, hepatic encephalopathy).
  * Presence of ≥F2 liver fibrosis if a patient has previously had a liver biopsy.
  * Have ALT or AST > upper limit of normal (ULN).
  * Total bilirubin levels > ULN; if documented Gilbert's Syndrome, total bilirubin >2 × ULN.
  * INR ≥1.2 at screening. If deemed appropriate by the investigator and/or prescribing physician, the patient may stop taking anticoagulants for an appropriate washout period or reversal with vitamin K and if indicated, a repeat INR within <1.2 would be acceptable.
  * Seropositive for hepatitis B (positive surface Ag).
  * Active hepatitis C by hepatitis C virus (HCV) antibody. If HCV antibody positive, must be HCV RNA polymerase chain reaction (PCR) negative.

Part B:

Inclusion Criteria:

* Males or females 18 - 70 years of age inclusive at the time of consent.
* Diagnosis of AATD and homozygous for the PiZZ mutation (confirmed by genetic testing).
* Evidence of METAVIR F1, F2, or F3 liver fibrosis based on a central read of a baseline liver biopsy during the screening period or a histological diagnosis made no more than 6 months before enrollment and stage confirmed by central read.
* A postbronchodilator FEV1 ≥40% of predicted at screening. (PFTs obtained within 1 year of signing the ICF may be used for eligibility.)

Exclusion Criteria:

* Lung or liver transplant or on waiting list for lung or liver transplant or status post lung volume reduction surgery.
* Clinical evidence of severe bronchiectasis as per the discretion of the investigator (eg, excessive sputum production or recurrent infections requiring antibiotic use [>4x/year])
* Previous diagnosis of liver cirrhosis or complications of cirrhosis (eg, varices, ascites, hepatic encephalopathy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Dose Exploration: Rates of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 2 years
  Numbers and percentages of patients reporting a given AE
Phase 2 Dose Expansion: Absolute blood levels of total AAT | 2 Years
  Absolute Levels of AAT over time

SECONDARY OUTCOMES:
Phase 1 Dose Exploration: Absolute blood levels of total AAT | 2 Years
  Absolute Levels of AAT over time
Phase 2 Dose Expansion: Rates of TEAEs and SAEs | 2 Years
  Numbers and percentages of patients reporting a given AE

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Beam Therapeutics
Locations (6):
- Australia (2):
  - Clinical Study Center, Adelaide
  - Clinical Study Center, Fitzroy
- Clinical Study Center, Leiden, Netherlands
- New Zealand (2):
  - Clinical Study Center, Auckland
  - Clinical Study Center, Hamilton
- Clinical Study Center, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No